CLINICAL TRIAL: NCT06036862
Title: A Prospective Clinical Study of Transanal and Transabdominal Combined Endoscopic Resection of Rectal Stenosis and Anal Reconstruction for Severe Rectal Anastomotic Stenosis
Brief Title: Utilization of Transanal Endoscopy in the Treatment of Anastomotic Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Principal investigator of the sixth affiliated hospital of Sun Yat-sen University, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU-TLCAS
Record Dates: First submitted 2023-08-10; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Anastomotic Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with severe rectal anastomotic stenosis (Experimental): Focusing on Patients with severe rectal anastomotic stenosis, espically long length and ultra lower firbrotic stenosis
  Interventions: Procedure: Transanal and transabdominal combined endoscopic resection of rectal stenosis and anal reconstruction

INTERVENTIONS:
Procedure: Transanal and transabdominal combined endoscopic resection of rectal stenosis and anal reconstruction — Laparoscopic or open surgery was selected according to the patient's condition, surgical history and surgeon's experience.According to the extent of the rectal stenosis, the proximal colon was dissected.A circular incision was made above the dentate line and the broken end was sutured. After the intestinal cavity was closed, a single port was inserted through the anus, and a transanal endoscopic platform was established after pneumoperitoneum infusion.The stenotic and scar segments were removed free upward.Through the pelvic cavity and into the abdominal cavity from the bottom up. The narrow rectum and proximal colon were pulled out of the anus through the anus, and the diseased bowel was removed. According to the distance of the remaining distal rectum, stapler or manual anastomosis or Bacon operation was selected.

SUMMARY:
Severe rectal anastomotic stenosis can not only cause intestinal obstruction, but also be accompanied by frequent defecation, which affects the quality of life, and patients face the outcome of permanent stoma or temporary stoma again. Traditional transabdominal resection and reconstruction of rectal anastomotic stenosis is more likely to occur due to unclear anatomical structure, dense scars around the intestinal canal, complications such as ureteral and urethral injury and massive presacral hemorrhage. In addition,41%of patients with anastomotic stenosis who underwent reoperation through abdominal surgery had anastomotic leakage again, and up to 30% of patients could not close the stoma. The advantages of transanal total mesorectal excision (taTME) using a transanal approach for total mesorectal excision in the treatment of middle and low rectal cancer with difficult pelvis have been demonstrated by our group. However, taTME has rarely been explored in the treatment of anastomotic stenosis. Our team retrospectively summarized the patients who underwent transabdominal transanal endoscopic resection and reconstruction of anastomotic stenosis (l-taTME), and initially demonstrated the safety and effectiveness of this surgical method, with a stoma closure rate of 90%. Although the advantages of l-taTME in the treatment of severe rectal anastomotic stenosis are obvious in theory and preliminary clinical practice, there is a lack of prospective studies. Therefore, the investigators plan to conduct a prospective clinical study to observe the safety and efficacy of l-taTME reconstruction surgery, and to provide high-level evidence-based medical basis for the selection of resection and reconstruction surgery for patients with rectal anastomotic stenosis.

DETAILED DESCRIPTION:
Colorectal cancer is the most common malignant tumor of the digestive tract. At present, surgery is still the main treatment for rectal cancer. Although stapler anastomosis improves the safety of surgical resection and reconstruction for middle and low rectal cancer, surgical complications, especially anastomotic leakage, are inevitable, especially for middle and low rectal cancer, where the incidence of anastomotic leakage reaches 8-11%. The outcome of anastomotic leakage will lead to anastomotic stenosis, especially in middle and low rectal cancer after neoadjuvant radiotherapy, and the incidence of anastomotic stenosis is as high as 3%-10%. Previous studies have suggested that anastomotic diameter < 20mm is considered as an anastomotic stenosis, and it has also been shown that an anastomotic diameter less than 1/3 of the original diameter of the intestinal lumen is considered as an anastomotic stenosis. Anastomotic stenosis can not only cause intestinal obstruction symptoms, such as abdominal distension and abdominal pain, but also be accompanied by frequent defecation, which affects the quality of life, and many patients face the outcome of permanent stoma or temporary stoma again.

Anastomotic stenosis is divided into membranous stenosis and tubular stenosis according to the degree of stenosis. For anastomotic membranous stenosis, endoscopic incision of the stenosis ring or balloon dilatation is the preferred method for the treatment of membranous stenosis. However, endoscopic scar incision and balloon dilation require repeated, multiple treatments to achieve long-term effectiveness, with the risk of perforation, pelvic infection, and bleeding. Balloon dilatation or scar incision has little effect on patients with low anastomosis position or tubular stenosis, and nearly 30% of patients need to undergo resection and reconstruction of the stenotic anastomosis. As anastomotic stenosis is often caused by anastomotic leakage, anastomotic ischemia, radiotherapy and chemotherapy, use of stapler, pelvic infection and low anastomosis, the anatomical structure is unclear, the scar around the bowel is dense, and complications such as ureteral and urethral injury and massive bleeding of presacral veins are more likely to occur during the resection and reconstruction of the stricture. Lefevre et al. reported 33 patients who underwent resection and reconstruction of transabdominal rectal anastomotic stenosis, and the incidence of perioperative complications was 54.5%, including anastomotic leakage of 18%（6/33） and postoperative intestinal obstruction of 12%. Genser et al. reported 50 patients with surgical treatment of anastomotic stenosis, of whom 12（24%） received intraoperative blood transfusion, with an average blood transfusion volume of 2.5 units. The incidence of intraoperative complications was 12%, including 5 cases of bladder injury and 1 case of splenectomy due to splenic injury due to unclear anatomical location. Westerduin et al. summarized 59 patients who underwent secondary surgery for anastomotic leakage and stenosis, and 41% of them had recurrent anastomotic leakage 14 months after surgery. During the follow-up of 27 months, only 66% of the patients regained intestinal continuity,24%of the patients received permanent colostomy, and 10% of the patients retained ileostomy.

Due to the difficulty of surgery, it is difficult to remove the scar tissue around the anastomosis in the traditional abdominal resection and reconstruction surgery. The new rectorectum cannot be pulled out and anastomosed with the distal rectoanal canal again. After reluctant anastomosis, the incidence of anastomotic leakage is still high due to the high tension of rectorectum, and many patients have to accept permanent stoma. Transanal total mesorectal excision (taTME), which uses a transanal approach to perform total mesorectal excision, has been demonstrated by our team for the surgical treatment of middle and low rectal cancer with difficult pelvis. However, the use of taTME in the treatment of anastomotic stenosis is rarely explored at present. Our team first reported this surgical method in 2021. The investigators retrospectively summarized 17 patients who underwent resection and reconstruction of anastomotic stenosis by transabdominal transanal endoscopic surgery. The ileostomy or colostomy was closed in 15 patients, which proved the safety and effectiveness of this surgical method. Transabdominal transanal endoscopic resection and reconstruction surgery has obvious advantages in the treatment of patients with rectal anastomotic stenosis. First, it can accurately separate the narrow distal intestine, and transanal anastomosis of the substitute rectum and the distal rectoanal canal can be performed, which reduces the difficulty of reconstruction. Secondly, from the distal normal anorectal canal, it can enter the normal anatomical structure space, and the narrow scar segment can be completely resected by endoscopic magnification. At the same time, it can reduce the accidental injury of the surrounding normal tissue and significantly reduce the incidence of intraoperative complications. Finally, the mobilization of the left hemicolon and splenic flexure of the abdomen was completed laparoscopically, and the specimen was removed through the anus, which did not require additional abdominal incision and thus reduced trauma. Although the advantages of transanal transabdominal combined with laparoscopic resection and reconstruction in the treatment of severe rectal anastomotic stenosis are very obvious in theory and preliminary clinical practice, there is a lack of prospective studies.

For the above reasons, the investigators plan to conduct a prospective clinical study to observe the safety and efficacy of transanal laparoscopic resection and reconstruction in patients with rectal anastomotic stenosis, in order to improve the quality of life of patients with rectal anastomotic stenosis, and to provide high-level evidence-based medical basis for the selection of resection and reconstruction surgery for patients with rectal anastomotic stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-70 years old;
2. ECOG performance status score 0-2;
3. previous rectal resection;
4. patients diagnosed with middle and low rectal anastomotic tubular stenosis;
5. can tolerate general anesthesia;
6. The subjects and their family members, who could understand the study protocol and were willing to participate, signed the informed consent form.

Exclusion Criteria:

1. patients with acute intestinal obstruction, intestinal perforation or intestinal bleeding requiring emergency surgery;
2. severe pelvic adhesion and frozen pelvis;
3. patients with unstable primary tumors or combined with tumors at other sites;
4. previous history of left hemicolectomy;
5. ASA grade IV to V;
6. combined organ resection;
7. severe mental illness;
8. pregnant or lactating women;
9. severe cardiovascular disease, uncontrolled infection or other uncontrolled comorbidities;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Stoma recovery rate | 3 months after surgery
  whether the stoma recovery and restoration of bowel continuation

SECONDARY OUTCOMES:
incidence of postoperative anastomotic leakage | 1 month after surgery
  whether the occurence of anastomotic leakage
incidence of postoperative anastomotic bleeding | Duration of 7 days after surgery
  whether the occurence of anastomotic bleeding
Incidence of severe bowel dysfunction | 3 months after stoma recovery
  Low Anterior Resection Syndrome Score (0-20: No LARS 21-29: Minor LARS 30-42: Major LARS)
Incidence of severe bowel dysfunction | 6 months after stoma recovery
  Low Anterior Resection Syndrome Score (0-20: No LARS 21-29: Minor LARS 30-42: Major LARS)
Incidence of severe bowel dysfunction | 1 year after stoma recovery
  Low Anterior Resection Syndrome Score (0-20: No LARS 21-29: Minor LARS 30-42: Major LARS)
Incidence of severe bowel dysfunction | 2 years after stoma recovery
  Low Anterior Resection Syndrome Score (0-20: No LARS 21-29: Minor LARS 30-42: Major LARS)
Anorectal function | 1 year after stoma recovery
  Anorectal pressure Rectal sensory function Rectoanal reflex function
Anorectal function | 2 year after stoma recovery
  Anorectal pressure Rectal sensory function Rectoanal reflex function
bowel function | 3 months after stoma recovery
  Memorial Sloan-Kettering Cancer Center bowel function instrument
bowel function | 6 months after stoma recovery
  Memorial Sloan-Kettering Cancer Center bowel function instrument
bowel function | 1 year after stoma recovery
  Memorial Sloan-Kettering Cancer Center bowel function instrument
bowel function | 2 year after stoma recovery
  Memorial Sloan-Kettering Cancer Center bowel function instrument
Quality of life evaluation after stoma closure | 3 months
  European Organization for Research and Treatment of Cancer QLQ-C30 (0-100 0：poor 100:best)
Quality of life evaluation after stoma closure | 6 months
  European Organization for Research and Treatment of Cancer QLQ-C30 (0-100 0：poor 100:best)
Quality of life evaluation after stoma closure | 1 year
  European Organization for Research and Treatment of Cancer QLQ-C30 (0-100 0：poor 100:best)
Quality of life evaluation after stoma closure | 2 years
  European Organization for Research and Treatment of Cancer QLQ-C30 (0-100 0：poor 100:best)
Quality of life evaluation after stoma closure | 3 years
  European Organization for Research and Treatment of Cancer QLQ-C30 (0-100 0：poor 100:best)
Inraoperative condition | In the process of operation
  operation time and whether to convert to laparotomy
Perioperative recovery time | perioperative period
  Duration of analgesics in hours For the first time the exhaust time in hours Time to first defecation in hours Time to first fluid intake in hours Time to resume normal diet in hours Abdominal drainage tube removal time in days Catheter removal time in days Length of postoperative hospital stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sixth Affiliated Hospital of Sun yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Brenner H, Kloor M, Pox CP. Colorectal cancer. Lancet. 2014 Apr 26;383(9927):1490-1502. doi: 10.1016/S0140-6736(13)61649-9. Epub 2013 Nov 11. PMID 24225001
- [Background] Lu P, Fields AC, Vise AS, Shabat G, Irani JL, Bleday R, Goldberg JE, Melnitchouk N. Anatomic Distribution of Colorectal Adenocarcinoma in Young Patients. Dis Colon Rectum. 2019 Aug;62(8):920-924. doi: 10.1097/DCR.0000000000001422. PMID 31162374
- [Background] Moran BJ. Stapling instruments for intestinal anastomosis in colorectal surgery. Br J Surg. 1996 Jul;83(7):902-9. doi: 10.1002/bjs.1800830707. PMID 8813772
- [Background] Braunschmid T, Hartig N, Baumann L, Dauser B, Herbst F. Influence of multiple stapler firings used for rectal division on colorectal anastomotic leak rate. Surg Endosc. 2017 Dec;31(12):5318-5326. doi: 10.1007/s00464-017-5611-0. Epub 2017 Jun 20. PMID 28634627
- [Background] Lee SY, Kim CH, Kim YJ, Kim HR. Anastomotic stricture after ultralow anterior resection or intersphincteric resection for very low-lying rectal cancer. Surg Endosc. 2018 Feb;32(2):660-666. doi: 10.1007/s00464-017-5718-3. Epub 2017 Jul 19. PMID 28726144
- [Background] Fegiz G, Angelini L, Bezzi M. Rectal cancer: restorative surgery with the EEA stapling device. Int Surg. 1983 Jan-Mar;68(1):13-8. PMID 6853077
- [Background] Hughes DL, Cornish J, Morris C; LARRIS Trial Management Group. Functional outcome following rectal surgery-predisposing factors for low anterior resection syndrome. Int J Colorectal Dis. 2017 May;32(5):691-697. doi: 10.1007/s00384-017-2765-0. Epub 2017 Jan 27. PMID 28130593
- [Background] Bruns ERJ, Borstlap WA, van Duijvendijk P, van der Zaag-Loonen HJ, Buskens CJ, van Munster BC, Bemelman WA, Tanis PJ. The Association of Preoperative Anemia and the Postoperative Course and Oncological Outcome in Patients Undergoing Rectal Cancer Surgery: A Multicenter Snapshot Study. Dis Colon Rectum. 2019 Jul;62(7):823-831. doi: 10.1097/DCR.0000000000001360. PMID 31188183
- [Background] Garcea G, Sutton CD, Lloyd TD, Jameson J, Scott A, Kelly MJ. Management of benign rectal strictures: a review of present therapeutic procedures. Dis Colon Rectum. 2003 Nov;46(11):1451-60. doi: 10.1007/s10350-004-6792-x. PMID 14605561
- [Background] Artifon EL, Castano Llano R, Otoch JP, Tchekmedyian AJ. [Endoscopic dilation of the gastrointestinal tract]. Rev Gastroenterol Peru. 2015 Jan;35(1):45-61. Spanish. PMID 25875518
- [Background] Nguyen-Tang T, Huber O, Gervaz P, Dumonceau JM. Long-term quality of life after endoscopic dilation of strictured colorectal or colocolonic anastomoses. Surg Endosc. 2008 Jul;22(7):1660-6. doi: 10.1007/s00464-007-9679-9. Epub 2007 Dec 11. PMID 18074183
- [Background] Suchan KL, Muldner A, Manegold BC. Endoscopic treatment of postoperative colorectal anastomotic strictures. Surg Endosc. 2003 Jul;17(7):1110-3. doi: 10.1007/s00464-002-8926-3. Epub 2003 May 6. PMID 12728381
- [Background] Kawada K, Sakai Y. Preoperative, intraoperative and postoperative risk factors for anastomotic leakage after laparoscopic low anterior resection with double stapling technique anastomosis. World J Gastroenterol. 2016 Jul 7;22(25):5718-27. doi: 10.3748/wjg.v22.i25.5718. PMID 27433085
- [Background] Vignali A, Fazio VW, Lavery IC, Milsom JW, Church JM, Hull TL, Strong SA, Oakley JR. Factors associated with the occurrence of leaks in stapled rectal anastomoses: a review of 1,014 patients. J Am Coll Surg. 1997 Aug;185(2):105-13. doi: 10.1016/s1072-7515(97)00018-5. PMID 9249076
- [Background] Lefevre JH, Bretagnol F, Maggiori L, Ferron M, Alves A, Panis Y. Redo surgery for failed colorectal or coloanal anastomosis: a valuable surgical challenge. Surgery. 2011 Jan;149(1):65-71. doi: 10.1016/j.surg.2010.03.017. Epub 2010 May 7. PMID 20451231
- [Background] Genser L, Manceau G, Karoui M, Breton S, Brevart C, Rousseau G, Vaillant JC, Hannoun L. Postoperative and long-term outcomes after redo surgery for failed colorectal or coloanal anastomosis: retrospective analysis of 50 patients and review of the literature. Dis Colon Rectum. 2013 Jun;56(6):747-55. doi: 10.1097/DCR.0b013e3182853c44. PMID 23652749
- [Background] Westerduin E, Borstlap WAA, Musters GD, Westerterp M, van Geloven AAW, Tanis PJ, Wolthuis AM, Bemelman WA, D'Hoore A. Redo coloanal anastomosis for anastomotic leakage after low anterior resection for rectal cancer: an analysis of 59 cases. Colorectal Dis. 2018 Jan;20(1):35-43. doi: 10.1111/codi.13844. PMID 28795776
- [Background] Remzi FH, El Gazzaz G, Kiran RP, Kirat HT, Fazio VW. Outcomes following Turnbull-Cutait abdominoperineal pull-through compared with coloanal anastomosis. Br J Surg. 2009 Apr;96(4):424-9. doi: 10.1002/bjs.6458. PMID 19283735
- [Background] Liu H, Zeng Z, Zhang H, Wu M, Ma D, Wang Q, Xie M, Xu Q, Ouyang J, Xiao Y, Song Y, Feng B, Xu Q, Wang Y, Zhang Y, Hao Y, Luo S, Zhang X, Yang Z, Peng J, Wu X, Ren D, Huang M, Lan P, Tong W, Ren M, Wang J, Kang L; Chinese Transanal Endoscopic Surgery Collaborative (CTESC) Group. Morbidity, Mortality, and Pathologic Outcomes of Transanal Versus Laparoscopic Total Mesorectal Excision for Rectal Cancer Short-term Outcomes From a Multicenter Randomized Controlled Trial. Ann Surg. 2023 Jan 1;277(1):1-6. doi: 10.1097/SLA.0000000000005523. Epub 2022 Jul 11. PMID 35815886
- [Background] Luo S, Zhang X, Hou Y, Hu H, Dong J, Wang L, Kang L. Transanal and transabdominal combined endoscopic resection of rectal stenosis and anal reconstruction based on transanal endoscopic technique. Surg Endosc. 2021 Dec;35(12):6827-6835. doi: 10.1007/s00464-020-08188-x. Epub 2021 Jan 4. PMID 33398554